CLINICAL TRIAL: NCT03469999
Title: Effect of Single Event Multi Level Chemoneurolysis With Dysport on Energy Expenditure and Walking Efficiency
Brief Title: Effect of Dysport Injections on Energy Expenditure and Walking Efficiency in Children With Cerebral Palsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR1322
Record Dates: First submitted 2018-01-24; First posted 2018-03-19 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy
Keywords: Botulinum toxin A; Walking efficiency; Spasticity; Dysport; Pediatric
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dysport Injectable Product (Experimental): All participants will participate in baseline data collection of energy expenditure, gait analysis, and lower limb spasticity assessment. All participants will receive single event multi level chemoneurolysis with Dysport and will have repeat data collection at 4 weeks and 12 weeks post injection.
  Interventions: Drug: Dysport Injectable Product

INTERVENTIONS:
Drug: Dysport Injectable Product — Selected dose of medication will be determined by affected muscle(s), severity of spasticity, and the patient's body weight. We will follow the recommended total Dysport dose of 10-15 units/kg per limb, not to exceed 15 units/kg for unilateral lower limb, 30 units/kg for bilateral lower limb, or a total of 1000 units, whichever is lower in a given session.
  Other Names: Botulinum toxin A

SUMMARY:
This study aims to evaluate the efficacy of single event multi level chemoneurolysis with the abobotulinumtoxin A drug, Dysport®, on walking energy expenditure and gait in children with spastic diplegia cerebral palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the leading cause of disability in children, with the most widespread type of CP being spastic CP which negatively affects physical function. Specifically it is reported that there is an increase in energy expenditure and oxygen consumption in children with CP. Single event multi level chemoneurolysis with abobotulinumtoxinA has been found to be an effective treatment for patients with spasticity to reduce energy expenditure by increasing walking efficiency; however many of these studies have conflicting methodological approaches. Therefore this study aims to evaluate the single event multilevel chemoneurolysis with Dysport® on energy expenditure and gait in children with spastic diplegia CP.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5-17 years. Must be <18 prior to injection.
* >10 kilograms at screening and injection visits
* Diagnosis of spastic diplegia or mild- to moderate spastic quadriplegia Cerebral Palsy
* Gross Motor Function Classification System level: I, II, III
* Ability to ambulate independently without aid, equinus gait
* Absent of joint or bone deformities
* Eligible to receive single-event multi-level chemoneurolysis (SEMLC)
* Cooperative and tolerant to testing procedures during clinic screening
* Presence of spasticity in one or both legs
* Be on a stable dose and regimen if on any prescribed medication/s
* Parent must have signed written informed consent and the Patient Authorization for Use and Release of Health and Research Study Information

Exclusion Criteria:

* Ankle contractures no more than -10 degrees with the knee extended
* Hemiplegia
* Wheelchair dependent
* Received Botulinum toxin within previous 4 months
* Uncontrolled epilepsy or certain types of seizures
* Fracture in the study limb within previous 12 months
* Infection or skin disorder at planned injection site
* Shortness of breath or other respiratory issues
* Uncontrolled clinically significant medical condition
* Received phenol or alcohol block in the study limb within previous 6 months
* Surgery in the study limb within previous 12 months
* Serial casting within previous 12 months
* New physiotherapy and/or orthotic regimen <1 month before study start. (physiotherapy and/or orthotic regimen will be permitted if it began >1 month before study start and maintained throughout study)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heakyung Kim, MD, Principal Investigator — Columbia University Medical Center- Department of Rehabilitation
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dysport Injectable Product
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dysport Injectable Product
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 12
Gross Motor Function Classification System (GMFCS) Diagnosis [Count of Participants; unit: Participants] — The Gross Motor Function Classification System (GMFCS) looks at movements such as sitting, walking and use of mobility devices. Grading is based on physical examination and physician's asssessents of a patient's clinical presentation. Grading ranges from GMFCS Level I, which includes children who walk without limitations but with some degree of difficulty with speed, balance, and coordination, (better outcome), to GMFCS Level V, which includes children who are transported in a manual wheelchair and have difficulty in head/trunk control (worse outcome).
  Participants
    GMFCS I (Children walk at home, school, outdoors and in the community) | 2
    GMFCS II (Children walk in most settings and climb stairs holding onto a railing) | 7
    GMFCS III (Children walk using a hand-held mobility device in most indoor settings) | 2
    Unknown (not part of analysis) | 1

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Consumption (ml/kg/Min)
Description: Energy expenditure (oxygen consumption (VO2)) will be measured during the 6 minute walk test using a portable metabolic cart. The participants will use a 10 meter walkway to walk back and forth during the 6 minutes to coverage as much distance as possible. During this time they will be wearing a portable spirometric device that collects the oxygen consumption (VO2) per minute.
Time Frame: Baseline (1 week prior to injection), 4 weeks post injection, 12 weeks post injection
Population: All participants who received Dysport and had VO2 level measured at baseline, week 4 and week 12.
Measure: Mean (95% Confidence Interval); unit: ml/kg/min
Arm/Group | Dysport Injectable Product
Number analyzed (Participants) | 11
ml/kg/min
  Baseline (pre-injection) | 14.82 [12.76 to 16.88]
  4 Week | 16.75 [13.53 to 19.96]
  12 Week | 28.77 [9.33 to 48.21]

2. Secondary Outcome: Gait Velocity (cm/s)
Description: Gait analysis will be measured by the GaitMat system while the child walks on the mat back and forth for five trials.
Time Frame: Baseline (1 week prior to injection), 4 weeks post injection, 12 weeks post injection
Population: Only includes participants who received Dysport and had gait analyzed at baseline, week 4 and week 12.
Measure: Mean (95% Confidence Interval); unit: cm/sec
Arm/Group | Dysport Injectable Product
Number analyzed (Participants) | 11
cm/sec
  Baseline (pre-injection) | 84.86 [67.90 to 101.81]
  4 weeks | 92.84 [80.04 to 105.06]
  12 weeks | 87.11 [66.76 to 197.47]

3. Secondary Outcome: Muscle Spasticity Using MAS
Description: The Modified Ashworth Scale (MAS) measures muscle spasticity during passive stretching. Scores are on a 6-point scale and include 0, 1, 1+, 2, 3, and 4. Scores range from 0 (better outcome), which indicates no increase in muscle tone/muscle spasticity to a score of 4 (worse outcome), which indicates a rigid muscle or maximum spasticity. Each subscale is independently scored and not combined to create a composite score. When calculating the mean score, 1+ is equivalent to a value of 1.5.
Time Frame: Baseline (1 week prior to injection), 4 weeks post injection, 12 weeks post injection
Population: Only includes participants who received Dysport and completed the MAS at baseline, week 4 and week 12.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dysport Injectable Product
Number analyzed (Participants) | 11
score on a scale
  MAS R Hip Adduction Baseline | 1.71 [1.26 to 2.17]
  MAS R Hip Adduction 4 week | 1.29 [0.83 to 1.74]
  MAS R Hip Adduction 12 week | 1.17 [0.38 to 1.96]
  MAS L Hip Adduction Baseline | 1.71 [1.26 to 2.17]
  MAS L Hip Adduction 4 week | 1.14 [0.79 to 1.49]
  MAS L Hip Adduction 12 week | 1.17 [0.38 to 1.96]
  MAS R Knee Flexion Baseline | 2.11 [1.65 to 2.57]
  MAS R knee Flexion 4 week | 1.44 [1.04 to 1.85]
  MAS R Knee Flexion 12 week | 1.89 [1.43 to 2.35]
  MAS L Knee Flexion Baseline | 1.89 [1.43 to 2.35]
  MAS L Knee Flexion 4 week | 1.78 [1.27 to 2.29]
  MAS L Knee Flexion 12 week | 1.78 [1.14 to 2.42]
  MAS R Dorsiflexion Baseline | 2.33 [1.95 to 2.72]
  MAS R Dorsiflexion 4 week | 1.89 [1.63 to 2.15]
  MAS R Dorsiflexion 12 week | 2.38 [1.94 to 2.81]
  MAS L Dorsiflexion Baseline | 2.11 [1.30 to 2.92]
  MAS L Dorsiflexion 4 week | 1.89 [1.43 to 2.35]
  MAS L dorsiflexion 12 week | 2.63 [1.86 to 3.39]

4. Secondary Outcome: Muscle Spasticity Using MTS
Description: The Modified Tardieu Scale (MTS) measures muscle spasticity during a passive stretch at both slow and fast speeds. Scores range from 0, which indicates no resistance throughout the course of the passive movement (better outcome), to 5, which indicates that the joint is immovable (worse outcome). The first measure determines the maximum range of motion of a target muscle group in degrees and the second measure determines the angle where muscle resistance is felt during a rapid velocity stretch, recorded in degrees. The total score is calculated by subtracting measure one from measure two. A greater difference between measures indicates less muscle spasticity. The Modified Tardieu Scale will be performed in the hamstrings, gastrocnemius, and soleus muscles.
Time Frame: Baseline (1 week prior to injection), 4 weeks post injection, 12 weeks post injection
Population: Data was not collected for any of the participants.
Groups:
- Dysport Injectable Product: All participants will participate in baseline data collection of energy expenditure, gait analysis, and lower limb spasticity assessment. All participants will receive single event multi level chemoneurolysis with Dysport and will have repeat data collection at 4 weeks and 12 weeks post injection.
  Selected dose of medication will be determined by affected muscle(s), severity of spasticity, and the patient's body weight. We will follow the recommended total Dysport dose of 10-15 units/kg per limb, not to exceed 15 units/kg for unilateral lower limb, 30 units/kg for bilateral lower limb, or a total of 1000 units, whichever is lower in a given session.
  Data was not analyzed
Arm/Group | Dysport Injectable Product
Number analyzed (Participants) | 0

5. Secondary Outcome: Score on the Cerebral Palsy Quality of Life (CP QOL) Questionnaire
Description: The Cerebral Palsy Quality of Life (CP QOL) Questionnaire consists of 66 items ranging from 1 to 9 with a lower score indicating a higher quality of life. The total score will be calculated as well as an individual score for the seven subscale domains: Social well-being and acceptance, functioning, Participation and physical health, Emotional well-being, Access to services, pain and feeling about disability, and family health. Scoring involves 2 steps. First, items are transformed to a scale with a possible range of 0-100. The scores are recoded as follows 1 to 0, 2 to 12.5, 3 to 25, 4 to 37.5, 5 to 50, 6 to 6.2, 7 to 75, 8 to 87.5, 9 to 100. Then the algebraic mean of item values is computed from the composite score for each domain. Once rescored, the final score ranges from 0 to 100, with 0 indicating a worse outcome.
Time Frame: Baseline (1 week prior to injection), 4 weeks post injection, 12 weeks post injection
Population: Data was not collected for any of the participants.
Arm/Group | Dysport Injectable Product
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Each participant was followed for up to 12 weeks post-injection for occurrence of any adverse events, serious adverse events and/or death. Adverse event data was collected over a period of approximately 1 year and 1 month, from December 12, 2018 to January 29, 2020.
Groups:
- Dysport Injectable Product: All participants will participate in baseline data collection of energy expenditure, gait analysis, and lower limb spasticity assessment. All participants will receive single event multi level chemoneurolysis with Dysport and will have repeat data collection at 4 weeks and 12 weeks post injection.
  Dysport Injectable Product: All participants will receive Dysport injection at multi levels in the spastic lower limb(s).
Arm/Group | Dysport Injectable Product
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT03469999/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03469999/ICF_001.pdf